CLINICAL TRIAL: NCT00404001
Title: A Phase 2, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Range-Finding Study of the Safety and Efficacy of Orally Administered MD-0727 in Patients With Primary Hypercholesterolemia
Brief Title: Study of Oral MD-0727 Administered to Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-104-201
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2007-09

CONDITIONS: Hypercholesterolemia
Keywords: Microbia; MD-0727; Primary Hypercholesterolemia; Hypercholesterolemia; Hyperlipidemia; Dyslipidemia; Cholesterol; LDL
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MD-0727

SUMMARY:
The primary objectives of this study are to evaluate the safety of MD-0727 in patients with primary hypercholesterolemia and to determine the low density lipoprotein cholesterol (LDL-C) lowering effect and dose-response of MD-0727 in patients with primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or non-pregnant, non-breastfeeding female, at least 18 years of age
* Patient must agree to use contraception and/or birth control if sexually active
* Patient may not be on lipid-lowering therapies at least 6 weeks prior to study and must have a fasting LDL-C 130 mg/dl or greater at Screening
* Patient must have an average of two fasting LDL-C measures greater than/equal to 130 mg/dl but less than/equal to 210 mg/dl with a difference in the two measures less than/equal to 15%. Patient may not have a fasting serum triglyceride less than 300 mg/dl during Pre-treatment Period
* Patient's BMI must be greater than/equal to 18.5 but less than 35.0 at Screening
* Patient must complete a physical exam, 12-lead ECG, and other laboratory tests (including pregnancy test) with no clinically-significant findings prior to the first dose of study medication
* Patient agrees to comply with the TLC diet
* Patient completes a 6-week washout of previous lipid-lowering medication including over-the-counter products

Exclusion Criteria:

* Patient has a medical condition that is prohibited per protocol or a condition that the Investigator believes may limit the patient's ability to participate in the study
* Patient has a TSH level >1.5 X the upper limit of normal
* Patient has history of cardiovascular or coronary artery disease, uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, or patient has history of NYHA Class III or IV congestive heart failure
* Patient is diabetic or presents with fasting blood glucose greater than/equal to 126 mg/dl at any time prior to randomization
* Patient has uncontrolled hypertension with a systolic blood pressure greater than/equal to 180 mm Hg or diastolic blood pressure greater than/equal to 110 mmg Hg at two study visits prior to the first dose of study medication
* Patient has a 10-year CHD risk of > 20%
* Patient has ALT or AST > 1.5 X the upper limit of normal prior to randomization
* Patient has a history of alcohol or drug abuse within 12 months of Screening
* Patient has used a prohibited medication (per protocol) during the 14-day Pre-treatment Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C)

SECONDARY OUTCOMES:
Total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Microbia Medical Affairs, Study Director — Microbia, Inc.
Locations (20):
- United States (20):
  - Microbia Investigational Site, Birmingham, Alabama
  - Microbia Investigational Site, Los Angeles, California
  - Microbia Investigational Site, Walnut Creek, California
  - Microbia Investigational Site, New Port Richey, Florida
  - Microbia Investigational Site, Chicago, Illinois
  - Microbia Investigational Site, Indianapolis, Indiana
  - Microbia Investigational Site, Overland, Kansas
  - Microbia Investigational Site, Louisville, Kentucky
  - Microbia Investigational Site, Edina, Minnesota
  - Microbia Investigational Site, Kansas City, Missouri
  - Microbia Investigational Site, Statesville, North Carolina
  - Microbia Investigational Site, Winston-Salem, North Carolina
  - Microbia Investigational Site, Cincinnati, Ohio
  - Microbia Investigational Site, Marion, Ohio
  - Microbia Investigational Site, Charleston, South Carolina
  - Microbia Investigational Site, Bristol, Tennessee
  - Microbia Investigational Site, San Antonio, Texas
  - Microbia Investigational Site, Richmond, Virginia
  - Microbia Investigational Site, Lakewood, Washington
  - Microbia Investigational Site, Olympia, Washington